CLINICAL TRIAL: NCT03405311
Title: 3D Ultrasound-guided Labor Epidural Analgesia in the Morbid Obese Parturient: A Randomized Control Trial
Brief Title: 3D Ultrasound-guided Labor Epidural Analgesia in the Morbid Obese Parturient
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study device is not working, and there is no funding available to purchase or rent a new one.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-0286
Record Dates: First submitted 2018-01-02; First posted 2018-01-23 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Obesity, Morbid; Pregnancy; Pain
Keywords: Labor analgesia; Ultrasound; Obesity, Morbid; Pregnancy; Labor Epidural Analgesia
MeSH Terms: conditions — Obesity, Morbid; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Palpation (Active Comparator): The control group (Group 2: Epidural) will receive the 'Blind/standard approach', which is the current standard of care using palpation in administering labor epidural analgesia. Additionally, an anesthesiologist will scan patient's back with Accuro device in turn off mode.
  Interventions: Other: Palpation
- Rivanna Accuro 3D Ultrasound Device (Experimental): The treatment group (Group 1: Ultrasound and Epidural) will receive epidural analgesia using ultrasound pre-procedural scan with the ACCURO device.
  Interventions: Device: Rivanna Accuro 3D Ultrasound Device

INTERVENTIONS:
Device: Rivanna Accuro 3D Ultrasound Device — The treatment group (Group 1: Ultrasound and Epidural) will receive epidural analgesia using ultrasound pre-procedural scan with the ACCURO device
  Arms: Rivanna Accuro 3D Ultrasound Device
Other: Palpation — The control group (Group 2: Epidural) will receive the 'Blind approach/palpation', which is using palpation in administering labor epidural analgesia. Additionally, anesthesiologist will scan patient's back with Accuro device in turned off mode
  Arms: Palpation

SUMMARY:
This study will be a randomized control study, with the objective to evaluate epidural analgesia success rates between the two methods (Blind Approach versus Accuro Device).

DETAILED DESCRIPTION:
Worldwide obesity has become an epidemic. The obstetrical population is no exception. This made more challenging for anesthesiologists on labor and delivery units to administer epidural analgesia. According to the World Health Organization, more than 30% of U.S. adults are obese with a body mass index (BMI; in kg/m2) ≥ 30. Recent data has shown that increased BMI has been associated with increased neuraxial analgesic failure and difficulty with prolonged epidural placement time.

The 'Blind approach' is the current standard of care in administering neuraxial anesthesia. The physician palpates the patient's spinal bony landmarks; the needle is placed in relation to identified landmarks and inserted until loss of resistance is felt. In the obese population, the success rates are as low as 68%. Recently the FDA has approved a handheld device "The Accuro" as an adjunct for neuraxial analgesia (Rivanna Medical, LLC). It consists of a three-dimensional ultrasound device. By utilizing sound waves it constructs three-dimensional images of the spinal column, allowing the physician to better see the spine in order to perform spinal/epidural anesthesia.

Hypothesize that this device will enable clinicians to assess epidural spaces for epidural needle placement compared with the traditional Blind approach in the morbidly obese parturient.

This study will be a randomized control study, with the objective to evaluate epidural analgesia success rates between the two methods (Blind Approach versus Accuro Device). Also, will determine if ultrasound based landmarks would reduce the needle tract and thereby reduced the amount of post-procedure pain at the insertion site in the peripartum period by using the algometer.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status class I, II, or III.
* Term pregnancy.
* Requesting epidural analgesia for anticipated vaginal delivery.
* BMI>or = 40.

Exclusion Criteria:

* Contraindication for epidural analgesia
* Inability to adequately understand the consent form.
* Incarcerated patients.
* Patients with known spinal deformities.
* Allergies to ultrasound gel.
* Allergies to local anesthetics

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Number of needle insertion attempts and redirections | Beginning of needle insertion till catheter placement-15 minutes
  An epidural insertion attempt will be defined as advancement of the needle in an effort to enter the epidural space; a needle requiring withdrawal for redirection or reinsertion through the skin/another skin puncture will be counted as an additional attempt
Successful epidural catheter placement | Within first 90 minutes following catheter placement
  Epidural failure-replacement will be recorded

SECONDARY OUTCOMES:
Procedural difficulty | Beginning of needle insertion till catheter placement-15 minutes
  Procedural difficulty will be rated by the performing anesthesiologist on a 10-point Likert scale from one (easy) to ten (extremely difficult).
Needle depth | Beginning of needle insertion till catheter placement-15 minutes
  We will also record thouy needle depth from skin and measured depth by ultrasound.
Pressure pain thresholds and pain scores | Before epidural placement and hospital discharge up to 3 days
  Pressure pain thresholds will be obtained immediately prior to the epidural placement. The force that the patient will be indicated uncomfortable will be recorded. Each intervertebral level will be measured once. The PPT will be measured the next day after the discontinuation of the epidural.Twenty-four hours post-partum, pain with analgesia during labor was assessed using the Numerical Rating Scale (NRS).
Complications | Within 30 days of admission
  Any complications related to the epidural will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Rovnat Babazade, MD, Principal Investigator — The University of Texas Medical Branch
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States

REFERENCES:
- See also: 510(k) clearance for the Rivanna Accuro ultrasound device — https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm?ID=K132736